CLINICAL TRIAL: NCT01135407
Title: Role of the Cortico-basal Ganglia Loops in Visual Attention: Effects of Dopaminergic and Subthalamic Nucleus Stimulation in Parkinson's Disease
Brief Title: Visual Selective Attention in Parkinson's Disease
Acronym: VSA-PD
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: POLLAK Pierre, Professor of Neurology, Unité des Troubles du Mouvement, Clinique de Neurologie, Grenoble University Hospital
Other Study IDs: 0914
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-06

CONDITIONS: Visual Attention in Parkinson's Disease
Keywords: Parkinson's disease; Deep brain stimulation; Subthalamic nucleus; Levodopa; Selective visual attention; Basal ganglia diseases
MeSH Terms: conditions — Parkinson Disease; Basal Ganglia Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- group #1: Parkinson's disease patients at a disease's stage characterized by motor complications
  Interventions: Other: Recording during computerized tests
- group #2: Parkinson's disease patients treated by subthalamic nucleus deep brain stimulation.
  Interventions: Other: Recording during computerized tests
- group #3: healthy controls
  Interventions: Other: Recording during computerized tests

INTERVENTIONS:
Other: Recording during computerized tests — Patients will perform more than one experimental session. In each experimental session 3 computerized tasks, which are suitable to study visual attention, decision making and motor performances will be presented. During these tests, participants have to responds the most quickly and accurately possible to the appearance on a computer display of a predetermined target stimuli, presented alone or in an array of signals.
  The computerized tests are administered in two different conditions of medication: with or without dopaminergic treatment, corresponding to two different experimental sessions.
  Groups: group #1
Other: Recording during computerized tests — Patients will perform more than one experimental session. In each experimental session 3 computerized tasks, which are suitable to study visual attention, decision making and motor performances will be presented. During these tests, participants have to responds the most quickly and accurately possible to the appearance on a computer display of a predetermined target stimuli, presented alone or in an array of signals. The computerized tests are administered in three different sets of electrical (without stimulation, or selective stimulation of the sensorimotor or associative/limbic part of the subthalamic nucleus) stimulation, corresponding to three different experimental sessions.
  Groups: group #2
Other: Recording during computerized tests — Participants will perform more than one experimental session. In each experimental session 3 computerized tasks, which are suitable to study visual attention, decision making and motor performances will be presented. During these tests, participants have to responds the most quickly and accurately possible to the appearance on a computer display of a predetermined target stimuli, presented alone or in an array of signals.The computerized tests are administered twice (in two different experimental sessions) to verify the performance repeatability.
  Groups: group #3

SUMMARY:
Parkinson's disease (PD), which is generally considered to be a motor disorder, is now known to be accompanied in many instances by a variety of cognitive defects. This can be explained considering that PD is a neurodegenerative and progressive disorder of the basal ganglia system, which works modulating not only motor, but also cognitive and emotional behaviours.

Concerning this, some studies suggest that non-demented PD patients may suffer from a voluntary selective visual attention orienting deficit, showing a reduced skill in focusing upon one target, and may be easily distracted from irrelevant but salient stimuli, with a consequent negative impact on their physical health, social interactions and quality of life.

Up to now, the evidence of the role of the basal-ganglia system in modulating visual attention functions is poor and indirect and the effects of dopaminergic and subthalamic nucleus (STN) stimulation (two usual and effective treatments in PD) on attention performances are controversial.

The main objectives of the project are: 1) to assess the visual selective attention as well as the distractibility in PD patients; 2) to study the effects of patient's usual antiparkinsonian treatments, that is dopaminergic and STN stimulation, on visual attention performances.

Secondly, from a clinical and neurophysiologic point of view, the investigators want to study the respective role of the dopaminergic pathways and the sensorimotor and associative/limbic cortico-basal ganglia loops passing across the STN in the visual attention performances.

To precisely answer the objectives of the protocol, the investigators will record the performances of participants during the administration of 3 computerized tests, which are suitable to study visual attention, decision making and motor performances.

The investigators will compare the performances on the computerized tests of two groups of PD patients, one evaluated in different sets of electrical (without stimulation, or selective stimulation of the sensorimotor or associative/limbic part of the STN) stimulation, the other in different conditions of medication (with or without dopaminergic treatment) with those of a group of healthy subjects.

DETAILED DESCRIPTION:
Study Model: parallel-groups study. Three groups of subjects will be enrolled for the study: 2 groups of PD patients (see for details the section groups/cohorts), and a group of healthy controls.

ELIGIBILITY:
PD patients and healthy controls will be matched for age, sex, and education. PD patients: group #1 e group #2

Inclusion Criteria:

* Idiopathic Parkinson's Disease at a disease's stage characterized by motor complications
* Able to tolerate a prolonged condition without medication
* Levodopa response > 30% (for group #1)
* Self-declared normal or corrected to normal vision
* At least one contact lead in the sensorimotor part and another contact in the associativelimbic part of the STN (for group #2).
* Patients with a healthy social security affiliation
* Able to give and sign the informed consent

Exclusion Criteria:

* Patients under guardianship, interdicted, or under administrative measures and legal constraints
* Fertile women not using adequate contraceptive methods
* Women who are pregnant or breast feeding
* Severe cognitive impairment
* Severe frontal executive functions impairment
* Actual psychotic disorders
* Major depression
* Motivation impairment
* Any medical or psychological problems which may interfere with a smooth conduction of the study protocol
* Significant deficiency in red-green color discrimination
* Drug or alcohol addiction

Healthy controls: group #3

Inclusion Criteria:

* Self-declared neurologically healthy subjects,
* Self-declared normal or corrected to normal vision
* No psychotropic or neurotrophic drugs intake
* Subjects with a healthy social security affiliation
* Able to give and sign the informed consent

Exclusion Criteria:

* Patients under guardianship, interdicted, or under administrative measures and legal constraints
* Fertile women not using adequate contraceptive methods
* Women who are pregnant or breast feeding
* Severe cognitive impairment
* Severe frontal executive functions impairment
* Actual psychotic disorders
* Major depression
* Motivation impairment
* Any medical or psychological problems which may interfere with a smooth conduction of the study protocol
* Significant deficiency in red-green color discrimination
* Drug or alcohol addiction

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients will be selected among those regularly treated in the Centres that take part to the study. Healthy controls will be selected among patient family circle, and the staff of the Centres where the research takes place.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
reaction time in trials of the computerized tests | 1 hour for each experimental session. All participants will perform more than one experimental session, on different days within the same week
  Reaction times is recorded during one hour sessions for each patient/control subject (for more details see the Intervention Section)

SECONDARY OUTCOMES:
responses accuracy in trials of the computerized tests | 1 hour for each experimental session. All participants will perform more than one experimental session, on different days within the same week
  responses accuracy is recorded during one hour sessions for each patient/control subject (for more details see the Intervention Section)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre POLLAK, Professor, Principal Investigator — Unité des Troubles du Mouvement, Clinique de Neurologie, Grenoble University Hospital
Locations (1):
- Unité des Troubles du Mouvement, Clinique de Neurologie, Grenoble University Hospital, Grenoble, France